CLINICAL TRIAL: NCT05721976
Title: Pilot Study of a Multigenerational Digital Lifestyle Intervention for Hispanic Female Cancer Survivors and Their Families
Brief Title: With Love, Grandma ("Con Cariño, Abuelita") Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami Sylvester Comprehensive Cancer Center (Other)
Collaborators: The V Foundation for Cancer Research (Other)
Responsible Party: Principal Investigator, Sara StGeorge, Assistant Professor of Public Health Sciences, University of Miami Sylvester Comprehensive Cancer Center
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20201421; 2018-024 (Other Grant/Funding Number: V Foundation for Cancer Research)
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Cancer, Breast; Cancer, Uterus; Cancer, Ovary; Obesity; Activity, Motor; Diet, Healthy
Keywords: Hispanic; family; digital health; cancer survivorship; physical activity; nutrition
MeSH Terms: conditions — Breast Neoplasms; Uterine Neoplasms; Ovarian Neoplasms; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Love, Grandma ("Con Cariño, Abuelita") Group (Experimental): Cancer survivor-Daughter dyads randomized to the With Love, Grandma ("Con Cariño, Abuelita") group will access a digital lifestyle program that includes 8 modules of didactic, behavioral, and family communication/parenting/grandparenting content from smartphones over the course of 10-12 weeks.
  Interventions: Behavioral: With Love, Grandma ("Con Cariño, Abuelita")
- Control Group (No Intervention): This group is intended to reflect typical services cancer survivors and family members receive from healthcare providers.

INTERVENTIONS:
Behavioral: With Love, Grandma ("Con Cariño, Abuelita") — Cancer survivor-Daughter dyads will log in to a secured website to access intervention content over a period of 10-12 weeks. The intervention will be delivered primarily through smartphones and will include 8 modules with didactic content on healthy lifestyle behaviors for cancer prevention and control, family behavior change content for setting weekly goals and self-monitoring health behaviors, and family communication and positive parenting/grandparenting content, all of which were developed in accordance with participant feedback based on formative intervention development work. In addition, and to increase participant compliance/reduce attrition often observed in digital health interventions, human support ("supportive accountability") will be provided. Specifically, each family will be assigned a "coach" who will use video conferencing software to engage in weekly 15-30 minute sessions regarding the family's progress throughout the intervention period.
  Arms: With Love, Grandma ("Con Cariño, Abuelita") Group

SUMMARY:
The purpose of this study is to assess the feasibility, acceptability, and preliminary effects of a digital (web and mobile-phone-based) program to improve lifestyle behaviors (physical activity, dietary intake) among Hispanic female cancer survivors and adult daughters.

ELIGIBILITY:
Cancer Survivor Inclusion Criteria:

* Grandmother
* Self-identifies as Hispanic
* Diagnosis of breast cancer (stages I-III), endometrial or ovarian cancer (stages I-II)
* Completed active treatment (i.e., surgery, chemotherapy, and/or radiation)
* Body Mass Index (BMI) ≥ 25 (overweight range)
* Engages in <150 minutes/week of moderate physical activity
* English or Spanish speaking
* Owns a mobile device with internet access (e.g., smartphone, tablet)
* Lives in South Florida

Daughter of Cancer Survivor Inclusion Criteria:

* Adult daughter of the identified cancer survivor (21 years of age or older)
* Has at least 1 living child ages ≤16 years old
* Body Mass Index (BMI) ≥ 25 (overweight range) OR engages in <150 minutes/week of moderate physical activity
* English or Spanish speaking
* Owns a mobile device with internet access (e.g., smartphone, tablet)
* Lives in South Florida

Daughter of Cancer Survivor Exclusion Criteria:

* Has been diagnosed with distant metastatic cancer
* Has not completed active treatment (i.e., surgery, chemotherapy, and/or radiation)
* Has uncontrolled schizophrenia or bipolar disorder
* Has a preexisting medical condition that precludes unsupervised physical activity (e.g., severe orthopedic conditions,wheelchair bound).

Cancer Survivor Exclusion Criteria:

* Has uncontrolled schizophrenia or bipolar disorder
* Has a preexisting medical condition that precludes unsupervised physical activity (e.g., severe orthopedic conditions, wheelchair bound)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Percent of survivor-daughter dyads retained at post-intervention (feasibility) | Up to 3 months
  Calculated by percent of enrolled survivor-daughter dyads who completed post-intervention measures
Percent of modules completed by survivor-daughter dyads (acceptability) | Up to 3 months
  Calculated as number of modules completed (of 8 total modules) by survivors and daughters

SECONDARY OUTCOMES:
Change in survivor and daughter physical activity as reported in the International Physical Activity Questionnaire (IPAQ) | Baseline, Up to 3 months
  Participants will self-report walking and sitting time (hours and minutes per day) using three items from the IPAQ. Mean difference in total time spent walking and sitting will be calculated from these items. The result is not reported in scales. Higher scores indicate higher time spent walking and sitting in the last 7 days.
Change in survivor and daughter physical activity as measured by the Godin Leisure Time Exercise Questionnaire | Baseline, Up to 3 months
  Responses range from 0 - greater than 24, with 0 indicating no activity and a higher score indicating more activities (no maximum score).
Change in survivor and daughter fruit and vegetable intake as measured by the NCI All-Day Screener | Baseline, Up to 3 months
  Participants will self-report dietary intake using the NCI All-Day Screener for fruit and vegetables and the percentage of energy from fat and fiber. Mean difference in cup equivalents of fruits and vegetables will be calculated using a scoring algorithm developed by the National Cancer Institute

CONTACTS AND LOCATIONS:
Overall Officials: Sara M St. George, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No